CLINICAL TRIAL: NCT02743260
Title: Single Centre in Vivo Cocktail Phenotyping Study on OATP1B1, OCT1/2, MATE1/2K, OAT1/3, and P-gp Drug Transporters in Healthy Volunteers
Brief Title: Drug Transporter Interaction Study PHENTRA_2015_KPUK
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Cologne (Other)
Collaborators: Umm Al-Qura University (Other); Institute for Biomedical and Pharmaceutical Research (IBMP), Nürnberg-Heroldsberg, Germany (Unknown)
Responsible Party: Principal Investigator, Prof. Dr. Uwe Fuhr, Acting Director, Department of Pharmacology I, University of Cologne
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: PHENTRA_2015_KPUK
Record Dates: First submitted 2016-04-11; First posted 2016-04-19 (Estimated); Last update posted 2019-09-10 (Actual); Status verified 2019-09

CONDITIONS: Healthy
Keywords: phenotype; transporter; cocktail
MeSH Terms: interventions — pitavastatin; Metformin; Digoxin; adefovir; adefovir dipivoxil; Sitagliptin Phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- pitavastatin (OATP1B1) (Experimental): 2 mg pitavastatin single dose
  Interventions: Drug: pitavastatin
- metformin (MATE1, MATE2K, OCT1, OCT2) (Experimental): 500 mg metformin single dose
  Interventions: Drug: Metformin
- digoxin (intestinal & renal P-glycoprotein) (Experimental): 0.5 mg digoxin single dose
  Interventions: Drug: digoxin
- adefovir dipivoxil (OAT1) (Experimental): 10 mg adefovir dipivoxil single dose
  Interventions: Drug: Adefovir
- sitagliptin (OAT3) (Experimental): 100 mg sitagliptin single dose
  Interventions: Drug: sitagliptin
- cocktail (all substances) (Experimental): combination of all individual drugs at respective single doses
  Interventions: Drug: pitavastatin; Drug: Metformin; Drug: digoxin; Drug: Adefovir; Drug: sitagliptin

INTERVENTIONS:
Drug: pitavastatin
  Other Names: Livazo®
  Arms: cocktail (all substances); pitavastatin (OATP1B1)
Drug: Metformin
  Other Names: Metformin-CT®
  Arms: cocktail (all substances); metformin (MATE1, MATE2K, OCT1, OCT2)
Drug: digoxin
  Other Names: Digacin®
  Arms: cocktail (all substances); digoxin (intestinal & renal P-glycoprotein)
Drug: Adefovir
  Other Names: Hepsera®
  Arms: adefovir dipivoxil (OAT1); cocktail (all substances)
Drug: sitagliptin
  Other Names: Januvia®
  Arms: cocktail (all substances); sitagliptin (OAT3)

SUMMARY:
The objective of the present study is to contribute to establishing in vivo phenotyping procedures for organic anionic transporter polypeptide 1B1 (OATP1B1), organic cation transporters 1 and 2 (OCT1/2), multidrug and toxic compound extrusion transporters 1 and 2,kidney splice variant (MATE1/2K), organic anion transporters 1 and 3 (OAT1/3), and p-glycoprotein (P-gp) transporters via a cocktail approach. To this end, marker substrates for each of the respective transporters are administered as single doses in one period each and as a cocktail in one period to 24 healthy volunteers, and phenotyping metrics are derived from plasma and urine concentrations.

DETAILED DESCRIPTION:
Blood sampling: - 0:15 h pre-dose, 0:15, 0:30, 0:45, 1:00, 1:20, 1:40, 2:00, 2:20, 2:40, 3:00, 3:30, 4:00, 5:00, 6:00, 8:00, 12:00, 16:00, 24:00 hours post-dose

Urine Sampling: Pre-dose, 0-4 hours, 4-8 hours, 8-12 hours, 12-16 hours, 16-24 hours

Drug analysis: by liquid chromatography - tandem mass spectrometry (LC-MS/MS)

Pharmacokinetic Characteristics: Evaluation is carried out using standard noncompartmental characteristics including: area under the plasma concentration vs. time curve truncated at time t (AUC0-t), area under the plasma concentration vs. time curve extrapolated to infinity (AUC0-∞), peak plasma concentration (Cmax), time of occurrence of Cmax (tmax), apparent elimination half-life (t½), clearance over bioavailability (CL/F), renal clearance (CLr) and renal secretion. The evaluation may be completed by compartmental population pharmacokinetic approaches.

Statistical evaluation: Pharmacokinetic characteristics are compared for cocktail administration vs. individual administration by standard average bioequivalence assessment.

Safety, tolerability: Adverse events, laboratory and clinical parameters and vital signs will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian
* Body mass index (BMI) between and inclusive 18.5 and 30 kg/m2
* Willing and capable to confirm written consent prior to enrolment after ample information has been provided
* Normal findings in the medical history unless the principal investigator considers an abnormality to be clinically relevant.
* Considered to be healthy by the principal investigator on the basis of extensive pre-study screening-

Exclusion Criteria:

Standard for healthy volunteers, including:

* Female subjects only: positive results in pregnancy test
* Female subjects only: lactating women
* Female subjects only: subjects who do not use or do not agree to use appropriate contraceptive methods during the study as defined in Note for Guidance on Non-Clinical Safety Studies for the Conduct of Human Clinical Trials for Pharmaceuticals (CHMP/ICH/286/95 modification)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-04; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
organic anionic transporter polypeptide 1B1 (OATP1B1): Clearance over bioavailability (CL/F) of pitavastatin | 24 hours
  PK parameter
organic cation transporters 1 and 2 (OCT1/2), multidrug and toxic compound extrusion transporters 1 and 2,kidney splice variant (MATE1/2K): Renal clearance (CLr) of metformin | 24 hours
  PK parameter
intestinal p-glycoprotein (P-gp): Peak Plasma Concentration (Cmax) of digoxin | 24 hours
  PK parameter
renal p-glycoprotein (P-gp): Renal clearance (CLr) of digoxin: | 24 hours
  PK parameter
organic anion transporter 1 (OAT1): Renal clearance (CLr) of adefovir | 24 hours
  PK parameter
organic anion transporter 3 (OAT3): Renal clearance (CLr) of sitagliptin | 24 hours
  PK parameter

CONTACTS AND LOCATIONS:
Overall Officials: Uwe Fuhr, Prof. Dr., Principal Investigator — Department of Pharmacology I, University Hospital Cologne Cologne, NRW, Germany, 50931
Locations (1):
- Department of Pharmacology I, University Hospital Cologne, Cologne, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hsin CH, Stoffel MS, Gazzaz M, Schaeffeler E, Schwab M, Fuhr U, Taubert M. Combinations of common SNPs of the transporter gene ABCB1 influence apparent bioavailability, but not renal elimination of oral digoxin. Sci Rep. 2020 Jul 27;10(1):12457. doi: 10.1038/s41598-020-69326-y. PMID 32719417
- [Derived] Trueck C, Hsin CH, Scherf-Clavel O, Schaeffeler E, Lenssen R, Gazzaz M, Gersie M, Taubert M, Quasdorff M, Schwab M, Kinzig M, Sorgel F, Stoffel MS, Fuhr U. A Clinical Drug-Drug Interaction Study Assessing a Novel Drug Transporter Phenotyping Cocktail With Adefovir, Sitagliptin, Metformin, Pitavastatin, and Digoxin. Clin Pharmacol Ther. 2019 Dec;106(6):1398-1407. doi: 10.1002/cpt.1564. Epub 2019 Aug 12. PMID 31247117